CLINICAL TRIAL: NCT05790824
Title: Benefits of Spa Therapy in Saint-Lary Soulan for Knee Osteoarthritis
Acronym: LARYTHERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Patrick BLIN, Principal Investigator, University of Bordeaux
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A02899-32; 74119 (Other: Portail épidémiologie-France/Health Databases)
Record Dates: First submitted 2023-02-24; First posted 2023-03-30 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
Keywords: pain; spa therapy; functional disability
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Intervention Model Description: External comparison study between Larytherm cohort patients and Thermarthrose control patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spa therapy (Experimental): Protocol of spa therapy in rheumatology for 3 weeks
  Interventions: Other: Spa therapy

INTERVENTIONS:
Other: Spa therapy — The "RH2" rheumatology treatment protocol will propose treatments that can be carried out with water from the SL5 borehole and will be composed of:
  * 54 treatments among the following treatments:
    * Swimming pool, 15 minutes (code 201)
    * Bath with aerobath, 10 minutes (code 205)
    * Bath with immersion shower, 10 minutes (code 206)
    * Cataplasm in multiple local application, 10 minutes (code 408)
  * 18 sessions of mobilization pool, 15 minutes (code 601)

SUMMARY:
The hypothesis is that the use of spa therapy in Saint-Lary Soulan for knee osteoarthritis treatment would have a therapeutic effect on this pathology.

The main objective of this external comparison study is to evaluate the comparative effectiveness at 6 months of spa therapy in the Saint-Lary Soulan spa center on functional disability and pain (MCII: Minimal Clinical Important Improvement) in knee osteoarthritis compared to the control group of the Thermarthrose multicenter randomized clinical trial, receiving standard cares.

The patients included in the Larytherm cohort will undergo a three-week spa therapy in Saint-Lary Soulan with a follow-up of 6 months after the end of spa therapy.

DETAILED DESCRIPTION:
Knee osteoarthritis is a frequent disease with important consequences for quality of life of patients. In France, prevalence was estimated at 7.6% among subjects between 40-75 years old. The management of knee osteoarthritis is essentially based on lifestyle and dietary measures and the use of analgesic treatment. Spa treatments are also part of the overall management of this pathology.

In this context, the spa town Saint-Lary Soulan requests the approval of the " Rheumatology " therapeutic orientation for its new borehole water (SL5), which requires a study (Larytherm) conducted according to the criteria of the French Academy of Medicine.

Secondary objectives are to evaluate 6 months after spa therapy in Saint-Lary Soulan, the evolution of:

* Body Mass Index (BMI),
* knee pain due to knee osteoarthritis,
* functional impact,
* fatigue,
* physical activity,
* quality of life,
* consumption of analgesic treatments,
* the occurrence of episodes of joint effusion requiring puncture/infiltration,
* the occurrence of adverse events.

The patients will be identified by local physicians or through a local public communication campaign. The patients with criteria of eligibility will complete a self-reported questionnaire before the beginning of spa therapy, after the spa therapy and 6 months after the end of spa therapy, and the physicians practising at the spa center will complete a medical questionnaire at inclusion and after the spa therapy.

ELIGIBILITY:
Inclusion Criteria:

* painful knee due to knee osteoarthritis diagnosed for more than 6 months (confirmed by the general practitioner responsible for the identification of the patient) with at least three of the six clinical criteria defined by the American College of Rheumatology:

  * age > 50 years
  * morning stiffness lasting < 30 minutes
  * articular crepitation when moving the knee
  * globular knee with bony hypertrophy on physical examination
  * periarticular bone pain on physical examination
  * absence of local heat on palpation
* Visual Analogue Scale for the evaluation of pain felt over the last eight days with a score greater than or equal to 3/10
* affiliated or benefiting from a Social Security plan
* agreeing to participate in the study, having completed and signed the Patient's Free and Informed Consent Form

Exclusion Criteria:

* knee osteoarthritis limited to the patello-femoral joint
* at least one of the following diseases/conditions:

  * Contra-indications for the realization of spa therapy: evolving cancer, dementia, severe dermatosis, infectious state not stabilized, pregnancy, severe cardiac and respiratory insufficiency, phlebitis, inflammatory rheumatism, psychosis, acute spinal pain
  * Acute arthritis of septic or inflammatory origin
* an index knee arthroplasty within the last 6 months or a planned arthroplasty on the index knee within the next 6 months
* corticosteroids infiltration or viscosupplementation within the last 3 months
* spa therapy within the previous 6 months
* link with the staff of the Saint-Lary Soulan spa center or the physicians participating in the study (family, employee, etc.)
* language barrier (unable to read the information letter, complete the patient agreement form or self-questionnaires)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with Minimal Clinically Important Improvement (MCII) | 6 months after the end of spa therapy
  Improvement from baseline of at least 9.1 points on the Western Ontario and McMaster University osteoarthritis (WOMAC) index standardized functional subscale of 0-100 and/or at least 1.99 cm on the Visual Analogue Scale (VAS) for pain without knee surgery, at 6 months.
  WOMAC index (functional subscale): functional assessment index for knee osteoarthritis, exploring the daily function. The scoring system used for the answers to the questions is the Lickert scale with 5 possible answers (none = 0; minimal = 1; moderate = 2; severe = 3; extreme = 4).
  Visual Analogue Scale for the evaluation of knee osteoarthritis-related pain for the index knee experienced over the last eight days. The scale is presented as a 10 cm horizontal line, the left end (= 0 cm) corresponding to no pain and the right end (= 10 cm) to the maximum imaginable pain.
  This outcome will be evaluated in the Larytherm cohort and compared to the control group of the Thermarthrose study.

SECONDARY OUTCOMES:
Relative change from baseline in the WOMAC functional subscale index at the end of the spa therapy and at 6 months after the end of the spa therapy. | Baseline, end of spa therapy (week 3) and 6 months after the end of spa therapy
  WOMAC index (functional subscale): functional assessment index for knee osteoarthritis, exploring the daily function. The scoring system used for the answers to the questions is the Lickert scale with 5 possible answers (none = 0; minimal = 1; moderate = 2; severe = 3; extreme = 4).
Relative change from baseline in the WOMAC index (full questionnaire) at the end of the spa therapy and at 6 months after the end of the spa therapy. | Baseline, end of spa therapy (week 3) and 6 months after the end of spa therapy
  WOMAC index (full questionnaire): functional assessment index for knee osteoarthritis, exploring three areas of analysis: pain, stiffness and daily function. The scoring system used for the answers to the questions is the Lickert scale with 5 possible answers (none = 0; minimal = 1; moderate = 2; severe = 3; extreme = 4).
Relative change from baseline in the knee osteoarthritis pain measured by the Visual Analogue Scale (VAS) for pain at the end of the spa therapy and at 6 months after the end of the spa therapy. | Baseline, end of spa therapy (week 3) and 6 months after the end of the spa therapy
  Visual Analogue Scale for the evaluation of knee osteoarthritis-related pain for the index knee experienced over the last eight days. The scale is presented as a 10 cm horizontal line, the left end (= 0 cm) corresponding to no pain and the right end (= 10 cm) to the maximum imaginable pain.
Relative change from baseline in fatigue measured by the Visual Analogue Scale (VAS) for fatigue at the end of the spa therapy and at 6 months after the end of the spa therapy. | Baseline, end of spa therapy (week 3) and 6 months after the end of spa therapy
  Visual Analogue Scale for the evaluation of fatigue on the day of filling out the self-questionnaire.The scale is presented as a 10 cm horizontal line, the left end (= 0 cm) corresponding to no fatigue and the right end (= 10 cm) to the maximum imaginable fatigue.
Relative change from baseline in Lequesne's algo-functional index at the end of the spa therapy and at 6 months after the end of the spa therapy. | Baseline, end of spa therapy (week 3) and 6 months after the end of spa therapy
  Questionnaire to assess the functional abilities and discomfort experienced by patients with knee osteoarthritis. Each question is scored, and the final score is classified as follows: 0-4: modest disability, 5-7: moderate disability, 8-10 points: significant disability, 11-13 points: very significant disability, ≥14 points: unbearable extreme disability.
Relative change from baseline in quality of life measured with the 12-item Short-Form health survey (SF12) at the end of the spa therapy and at 6 months after the end of the spa therapy. | Baseline, end of spa therapy (week 3) and 6 months after the end of spa therapy
  Quality of life questionnaire exploring 8 dimensions of quality of life and calculating two Summary Psychological and Physical Scores, ranging from 0 (no quality of life) to 100 (maximum quality of life).
Relative change from baseline in BMI at 6 months after the end of the spa therapy. | Baseline and 6 months after the end of spa therapy
Consumption of analgesic treatments (analgesics, chondroprotective or anti-arthritic, intra-articular injections of corticoids and hyaluronic acid, physical treatments) with a patient self-questionnaire at baseline and 6 months after the spa therapy. | Baseline and 6 months after the end of spa therapy
  The patient self-questionnaire includes yes/no questions and pre-listed options.
Evolution from baseline of physical activity measured with the International Physical Activity Questionnaire (IPAQ-short version) at 6 months after the spa therapy. | Baseline and 6 months after the end of spa therapy
  Questionnaire for the assessment of physical activity performed for at least 10 minutes in a row during the last 7 days, including questions on heavy lifting. The score is expressed in metabolic equivalent task (MET-minutes/week) or categorically in 3 levels (low/moderate/high)
Occurrence of episodes of joint effusion requiring puncture/infiltration during the 6 months after spa therapy. | 6 months after the end of spa therapy
Occurrence of adverse events during spa therapy and the 6 months after spa therapy. | End of spa therapy (week 3) and 6 months after the end of spa therapy
Occurrence of work stoppages due to knee osteoarthritis during the 6 months after spa therapy. | 6 months after the end of spa therapy

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Blin, Principal Investigator — Bordeaux PharmacoEpi
Locations (1):
- Centre thermal de Saint-Lary Soulan, Saint-Lary-Soulan, France

REFERENCES:
- [Result] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131